CLINICAL TRIAL: NCT03456180
Title: Changes in Microvascular Perfusion During Blood Purification With Cytosorb® in Septic Shock
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Professor, Università Politecnica delle Marche
Other Study IDs: cyto2018
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Septic Shock
Keywords: septic shock; microcirculation; acute renal failure; renal replacement therapy; haemoadsorption
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Haemoadsorption with Cytosorb cartridge: patients with septic shock and acute renal failure requiring renal replacement therapy with the haemoadsorption cartridge Cytosorb
  Interventions: Device: Haemoadsorption with Cytosorb cartridge

INTERVENTIONS:
Device: Haemoadsorption with Cytosorb cartridge — microcirculatory monitoring in septic shock patients requiring renal replacement therapy for acute renal failure and haemoadsorption with Cytosorb cartridge

SUMMARY:
Sepsis is defined as a life-threatening event due to a dysregulated immune response to an host. Blood purification techniques may be considered as a therapeutic weapon to front sepsis and septic shock.

Haemoadsorption is one of the known blood purification technique that is employed in this study, and it is based on the principle that whole blood, contacting the surface of proper designed sorbent, would be cleared of certain substrates. With haemoadsorption it is possible to de-circulate from bloodstream high molecular weight substances, such as cytokines.In this study Cytosorb® cartridge, based on haemoadsorption principle is applied on septic patients, suffering for acute kidney failure, along with continuous veno-venous haemodialysis (CVVH-D).Microcirculation has a crucial role in the natural history of sepsis.

In this prospective observational non interventional study, 10 septic patients with an acute kidney failure that need CVVH are enrolled.

The primary endpoint of the study is to verify an improvement in the density of microcirculatory vessels and in the quality of blood flow after exposure to Cytosorb®. These two parameters are well described synthetically by the Perfused Vessel Density (PVD).

As secondary endpoints we also want to analyze the modification of microcirculation after haemoadsorption therapy: microvascular blood flow, described by the microvascular flow index (MFI) and peripheral tissue oxygen perfusion during Cytosorb® exposure using near infrared spectroscopy technique (NIRS)

DETAILED DESCRIPTION:
Introduction Sepsis is defined as a life-threatening event due to a dysregulated immune response to an infection. Blood purification techniques may be considered as a therapeutic weapon to front sepsis and septic shock.

The rationale of blood purification in sepsis is to modulate a dysregulated profile of immune response to the host in order to reduce tissue damage due to over production of pleiotropic pro-inflammatory cytokines.

Blood purification may also control elevated levels of anti-inflammatory cytokines that may lead to a down-modulation of immune system and immunoparalysis.

Haemoadsorption is one of the known blood purification technique that is employed in this study, and it is based on the principle that whole blood, contacting the surface of proper designed sorbent, would be cleared of certain substrates. With haemoadsorption it is possible to de-circulate from bloodstream high molecular weight substances, such as cytokines.

In this study Cytosorb® cartridge, based on haemoadsorption principle is applied on septic patients, suffering for acute kidney failure, along with continuous veno-venous haemodialysis (CVVH-D).

The immune system is involved in the pathogenesis of sepsis, but also the microcirculation has a crucial role in the natural history of this syndrome.

When a proinflammatory subset of cytokines is over-expressed, inducible nitric oxide synthase is activated and leads to an extra production on nitric oxide that results in a disrupted regulation of microvascular and capillary tone. The microcirculation plays a fundamental role to regulate gas, nutrients and metabolites exchange between bloodstream and cells. When microvascular perfusion is altered, tissue hypoxia may occur and result in organ dysfunction.

Microcirculation analysis can be performed at the bedside using a non-invasive video microscopy technique.

The primary endpoint of the study is to verify an improvement in the density of microcirculatory vessels and in the quality of blood flow after exposure to Cytosorb®. These two parameters are well described synthetically by the Perfused Vessel Density (PVD).

As secondary endpoints the investigators will analyze the modification of microcirculatory blood flow after haemoadsorption therapy. The microvascular blood flow, described by the microvascular flow index (MFI), is altered in sepsis. MFI values go from 0 to 3, where 0 means absence of flow, and 3 continuous blood flow. In septic shock MFI generally results to be inferior than 2.6, which is the cut off value between normal and altered MFI. Increasing value of MFI is a sign of microcirculation good response to therapy.

The investigators will also evaluate peripheral tissue oxygenation during Cytosorb exposure using near infrared spectroscopy (NIRS, Inspectra model 560 Hutchinson®). This technique evaluates microvascular perfusion on the thenar eminence muscle. A vascular occlusion test, that reproduces a stagnant ischemia condition, is performed to evaluate microvascular reactivity to an ischemia-reperfusion insult.

An improvement in tissue perfusion and microvascular reactivity is expected during the treatment.

Invasive haemodynamic monitoring will be performed using Picco2®. Changes in macro-haemodynamic parameters are expected in response to therapy.

The Sequential Organ Failure Assessment (SOFA) score will be calculated at the enrollment in this study and during the therapy.

Heart rate, SpO2, temperature, mean arterial pressure, arterial and central venous blood gas analyses will be collected during the study.

Materials and methods

In this prospective observational non interventional study, 10 septic patients with an acute kidney failure that need continuous veno-venous haemodialysis will be enrolled.

Prior to enrollment a formal informed consent is obtained. This study is approved by the local ethical committee.

Statistical analysis

The Kolmogorov-Smirnov test will be performed to define the normal or non-normal distribution of the variables. The ANOVA test for repeated measures with Bonferroni post hoc test or Dunn's post hoc test will be applied to evaluate differences over time. The Friedman test will be applied for not normally distributed data.

Blood sampling

At baseline (T0) participants will undergo arterial blood gas analysis to obtain the following values: arterial O2 tension (PaO2), arterial carbon dioxide tension, pH, base excess, lactate concentration, PaO2/FiO2 ratio, and central venous gas analysis to determine central venous O2 saturation.

The plasmatic concentration of the main pleiotropic cytokines will be measured, including interleukin (IL)1-beta, IL6, IL8, IL10, tumor necrosis factor-alpha.

After enrollment, these essay will be repeated at T1 (after 6h of exposure to Cytosorb®) and at T2 after 24h of therapy.

Routine blood cell count, clotting profile and leukocyte formula will be performed at baseline and at T2 along with proCalcitonine essay.

Microcirculation analysis

The investigators will analyse the microcirculation using sidestream dark field video microscopy technique applied to the sublingual mucosa, this technique is not invasive and painless.

In this study the investigators will use the Microscan by Microvision Medical (The Netherlands).

Three short videos of the microcirculation will be collected, captured in three different areas of the sublingual mucosa. These videos will be analysed using Automated Vascular Analysis (AVA 3.2 software, Microvision Medical, Amsterdam, NL). Microcirculation density is described by Total Vessel Density (TVD) and the De Backer score; microcirculation quality of flow is defined by the Microvascular flow index (MFI) and Percentage of Perfused Vessel (PPV). The Perfused Vessel Density (PVD) describes the density of well perfused vessel. Microcirculation analysis will be performed at T0, T1 and T2.

Tissue oxygenation

Tissue oxygenation will be assessed using near infrared spectroscopy (NIRS) applied on the thenar eminence muscle.

The device Inspectra® (Hutchinson model 560) measures the tissue oxygen saturation, and estimates the tissue haemoglobin content that is summarized in the tissue haemoglobin index (THI).

A vascular occlusion test will be performed, which simulates an ischemia-reperfusion condition of the tissue in order to evaluate microvascular reactivity.

A cuff is applied to the forearm and inflated at 300 mmHg in order to generate a stagnant ischemia. Inspectra screen generates a curve of desaturation named Downslope. When a value of tissue O2 saturation of 40% is reached, the occlusion cuff is deflated and the Inspector screen draws a curve of resaturation of the tissue, named Upslope. Upslope and Downslope values are measured. In the phase of resaturation an Hyperemia Area is obtained as tissue O2 saturation generally exceeds for a certain period of time the basal value. The hyperemia area is measured as an index of microvascular reactivity.

NIRS with a vascular occlusion test will be performed at T0, T1 and T2.

Haemodynamic monitoring

Each participant will undergo haemodynamic monitoring with transpulmonary thermodilution based devices (Picco2® by Pulsion and EV1000® by Edwards). Thermodilution based calibration are obtained ad basal time, at T1 and T2.

Vasopressor dose, haemodynamic parameters and SOFA score will be recorded at t0, t1, t2..

ELIGIBILITY:
Inclusion Criteria:

* age>18
* septic patients with acute kidney failure that need to undergo CHHV treatment.

Exclusion Criteria:

* hypersensitivity or allergy to the components of the cartridge
* pregnancy
* maxillary-facial trauma that prohibits mouth access and sublingual microcirculation evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with septic shock requiring renal replacement therapy for acute renal failure and undergoing haemoadsorption with Cytosorb cartridge
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
improvement in perfused vessel density | 24 hours
  improvement in perfusion of the sublingual microcirculation

SECONDARY OUTCOMES:
improvement in microvascular flow index | 6 hours and 24 hours
  improvement in microvascular blood flow quality
improvement in tissue oxygenation | 6 hours and 24 hours
  improvement in NIRS-derived parameters of tissue oxygenation and microvascular reactivity
improvement in perfused vessel density | 6 hours
  improvement in perfusion of the sublingual microcirculation

REFERENCES:
- [Background] Malacarne P, Stella A, Giudici D, Bertolini G. [Infection surveillance in intensive care units. Preliminary results of a multicenter GiViTI study in 71 Italian ICUs]. Minerva Anestesiol. 2004 May;70(5):321-8. Italian. PMID 15181412
- [Background] Suntharalingam G, Perry MR, Ward S, Brett SJ, Castello-Cortes A, Brunner MD, Panoskaltsis N. Cytokine storm in a phase 1 trial of the anti-CD28 monoclonal antibody TGN1412. N Engl J Med. 2006 Sep 7;355(10):1018-28. doi: 10.1056/NEJMoa063842. Epub 2006 Aug 14. PMID 16908486
- [Background] Hotchkiss RS, Coopersmith CM, McDunn JE, Ferguson TA. The sepsis seesaw: tilting toward immunosuppression. Nat Med. 2009 May;15(5):496-7. doi: 10.1038/nm0509-496. PMID 19424209
- [Background] Ronco C, Tetta C, Mariano F, Wratten ML, Bonello M, Bordoni V, Cardona X, Inguaggiato P, Pilotto L, d'Intini V, Bellomo R. Interpreting the mechanisms of continuous renal replacement therapy in sepsis: the peak concentration hypothesis. Artif Organs. 2003 Sep;27(9):792-801. doi: 10.1046/j.1525-1594.2003.07289.x. PMID 12940901
- [Background] Honore PM, Matson JR. Extracorporeal removal for sepsis: Acting at the tissue level--the beginning of a new era for this treatment modality in septic shock. Crit Care Med. 2004 Mar;32(3):896-7. doi: 10.1097/01.ccm.0000115262.31804.46. No abstract available. PMID 15090989
- [Background] Di Carlo JV, Alexander SR. Hemofiltration for cytokine-driven illnesses: the mediator delivery hypothesis. Int J Artif Organs. 2005 Aug;28(8):777-86. doi: 10.1177/039139880502800803. PMID 16211527
- [Background] Peng Z, Singbartl K, Simon P, Rimmele T, Bishop J, Clermont G, Kellum JA. Blood purification in sepsis: a new paradigm. Contrib Nephrol. 2010;165:322-328. doi: 10.1159/000313773. Epub 2010 Apr 20. PMID 20427984
- [Background] Cruz DN, Antonelli M, Fumagalli R, Foltran F, Brienza N, Donati A, Malcangi V, Petrini F, Volta G, Bobbio Pallavicini FM, Rottoli F, Giunta F, Ronco C. Early use of polymyxin B hemoperfusion in abdominal septic shock: the EUPHAS randomized controlled trial. JAMA. 2009 Jun 17;301(23):2445-52. doi: 10.1001/jama.2009.856. PMID 19531784
- [Background] Livigni S, Bertolini G, Rossi C, Ferrari F, Giardino M, Pozzato M, Remuzzi G; GiViTI: Gruppo Italiano per la Valutazione degli Interventi in Terapia Intensiva (Italian Group for the Evaluation of Interventions in Intensive Care Medicine) is an independent collaboration network of Italian Intensive Care units. Efficacy of coupled plasma filtration adsorption (CPFA) in patients with septic shock: a multicenter randomised controlled clinical trial. BMJ Open. 2014 Jan 8;4(1):e003536. doi: 10.1136/bmjopen-2013-003536. PMID 24401721
- [Background] Ince C. The microcirculation is the motor of sepsis. Crit Care. 2005;9 Suppl 4(Suppl 4):S13-9. doi: 10.1186/cc3753. Epub 2005 Aug 25. PMID 16168069
- [Background] Sakr Y, Dubois MJ, De Backer D, Creteur J, Vincent JL. Persistent microcirculatory alterations are associated with organ failure and death in patients with septic shock. Crit Care Med. 2004 Sep;32(9):1825-31. doi: 10.1097/01.ccm.0000138558.16257.3f. PMID 15343008
- [Background] Goedhart PT, Khalilzada M, Bezemer R, Merza J, Ince C. Sidestream Dark Field (SDF) imaging: a novel stroboscopic LED ring-based imaging modality for clinical assessment of the microcirculation. Opt Express. 2007 Nov 12;15(23):15101-14. doi: 10.1364/oe.15.015101. PMID 19550794
- [Background] Boushel R, Langberg H, Olesen J, Gonzales-Alonzo J, Bulow J, Kjaer M. Monitoring tissue oxygen availability with near infrared spectroscopy (NIRS) in health and disease. Scand J Med Sci Sports. 2001 Aug;11(4):213-22. doi: 10.1034/j.1600-0838.2001.110404.x. PMID 11476426
- [Background] De Backer D, Hollenberg S, Boerma C, Goedhart P, Buchele G, Ospina-Tascon G, Dobbe I, Ince C. How to evaluate the microcirculation: report of a round table conference. Crit Care. 2007;11(5):R101. doi: 10.1186/cc6118. PMID 17845716
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; International Sepsis Definitions Conference. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Intensive Care Med. 2003 Apr;29(4):530-8. doi: 10.1007/s00134-003-1662-x. Epub 2003 Mar 28. PMID 12664219